CLINICAL TRIAL: NCT01284985
Title: Short Term Follow-up of Patient Implanted With the Metatarso-Phalangeal Prosthesis METIS®
Status: Completed | Type: Observational
Sponsor: Integra LifeSciences Services (Industry)
Responsible Party: Sponsor
Other Study IDs: RECON-EMEA-05
Record Dates: First submitted 2011-01-26; First posted 2011-01-27 (Estimated); Last update posted 2014-09-11 (Estimated); Status verified 2014-09

CONDITIONS: Hallux Rigidus; Hallux Limitus; Hallux Valgus; Osteoarthritis; Rheumatoid Arthritis - Ankle and/or Foot
MeSH Terms: conditions — Hallux Rigidus; Hallux Limitus; Hallux Valgus; Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- METIS: Patient who has an indication of : Hallux Rigidus, Hallux Limitus with degenerative joint disease, Painful Hallux Valgus, Osteoarthritis, Rheumatoid arthritis, Post-traumatic arthritis and for which surgeon has recommended that a METIS® prosthesis be implanted.

SUMMARY:
The great toe is vital for normal, pain free ambulation. Decreased function associated with osteoarthritis of the first matatarsal phalangeal joint (MTP I) often called Hallux Rigidis or Hallux Limitus leading to a painful great toe. Patients experience pain during ambulation especially during the push-off phase of gait. When surgery is indicated four techniques are used for hallux rigidis; cheilectomie, resection arthroplasty, arthrodesis and implant surgery (1). Endoprostetic implants are relatively new. Silicone Implants like the arthroplasty developed by Swanson (2) resulted in foreign body reactions and periarticular bone loss. Subsequent implants, in particular the metallic hemi arthroplasty with or without polyethylene articulations, have been more successful (3). Still, implants are prone to wear of the material and show higher rates of loosening and infection compared to other techniques (4;5). In the last decades several new implants are described using two non cemented pressfit components, of titanium alloy or ceramic (6-9). Between 2001 and 2004 the investigators developed a new concept with instrumentation for exact alignment to prevent for wear with loosening of the implant on the long term. The implant has bone-conserving characteristics to enable arthrodesis as a salvage procedure. It is a completely modular two-component press fit titanium alloy implant with polyethylene insert that can be used as either for hemi-, total- or revision arthroplasty.

The purpose of this study is to have an overview of clinical status of the patient implanted with the METIS® prosthesis at short term (2 years of follow-up). The objective of this study is to evaluate the safety and efficacy of the Metatarso-Phalangeal prosthesis METIS® at short term follow up.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Have willingness to give his/her data transfer authorisation;
* has an indication of: Hallux Rigidus, Hallux Limitus with degenerative joint disease, Painful Hallux Valgus, Osteoarthritis, Rheumatoid arthritis, Post-traumatic arthritis, for which surgeon has recommended that a METIS® prosthesis be implanted

Exclusion Criteria:

* active infection or inflammation;
* excessive bone loss, bone deficiency or rapid joint destruction;
* suspected or documented metal allergy or intolerance;
* metatarsal head or phalangeal avascular necrosis;
* joint instability involving soft and fibrous tissue deficiency;
* severe metatarso-phalangeal axis deviation (Hallux Valgus angle > 20°);
* prior mental illness or patient demonstrates that their mental capacity may interfere with their ability to follow the study protocol;
* a previous joint replacement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject who has an indication of:
  * Hallux Rigidus;
  * Hallux Limitus with degenerative joint disease;
  * Painful Hallux Valgus;
  * Osteoarthritis;
  * Rheumatoid arthritis;
  * Post-traumatic arthritis. For which surgeon has recommended that a METIS® prosthesis be implanted
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2009-02; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
occurrence of device related complications | at 2 years

SECONDARY OUTCOMES:
improvement of the AOFAS Hallux Metatarsophalangeal-Interphalangeal Scale (HMIS) score (American Orthopaedic Foot and Ankle Society) | at 2 year
Device related complications | 1 year
AOFAS HMIS score | 1 year
Quality of Life score | overtime
X-ray evaluation | overtime

CONTACTS AND LOCATIONS:
Locations (4):
- Nemocnice Havlíčkův Brod, Havlíčkův Brod, Czechia
- Medisch Centrum Alkmaar, Alkmaar, Netherlands
- The Netcare and Linksfield Medical Centre, Johannesburg, South Africa
- Hospital clinico y provincial, Barcelona, Spain